CLINICAL TRIAL: NCT04382586
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled Study of Zanubrutinib Treatment in Patients Hospitalized for COVID-19 Infection and Pulmonary Distress
Brief Title: Covid-19 Infection and Pulmonary Distress Treatment With Zanubrutinib in Hospitalized Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-3111-219
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Pulmonary Complications; COVID-19
Keywords: Corona Virus; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — zanubrutinib; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zanubrutinib + Supportive Care (Experimental): Participants received zanubrutinib plus supportive care
  Interventions: Drug: Zanubrutinib; Drug: Supportive Care
- Placebo + Supportive Care (Active Comparator): Participants received placebo plus supportive care alone
  Interventions: Drug: Supportive Care; Drug: Placebo

INTERVENTIONS:
Drug: Zanubrutinib — 320 mg (4 x 80 mg) capsules administered orally once daily
  Other Names: BGB-3111; Brukinsa
  Arms: Zanubrutinib + Supportive Care
Drug: Supportive Care — Supportive care treatment was selected and administered as deemed appropriate by the study investigator
Drug: Placebo — Placebo to match zanubrutinib
  Arms: Placebo + Supportive Care

SUMMARY:
The primary objective of this study was to evaluate if the addition of zanubrutinib to supportive care increases the respiratory failure-free survival rate at Day 28 in participants hospitalized for Corona Virus Disease 2019 (COVID-19) and pulmonary distress not receiving mechanical ventilation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Hospitalization for COVID-19 infection
2. Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR)
3. Participant requires supplemental oxygen for pulmonary distress related to COVID-19 infection, and has been on supplemental oxygen for no more than 96 hours from time of screening

Key Exclusion Criteria:

1. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
2. On a Bruton's tyrosine kinase (BTK) inhibitor
3. Planned or concurrent use of a host modifiers/immune-based therapies or anti-CD20 monoclonal antibody treatment
4. Participants with prior of current hematologic malignancy or solid tumor malignancy with treatment within 6 months prior to study entry

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (10):
- United States (10):
  - St Jude Medical Center, Fullerton, California
  - Medstar Heath Research Institute Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - John D Archbold Memorial Hospital, Thomasville, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Brigham and Womens Hospital, Inc, Boston, Massachusetts
  - Rutgers University Hospital, Newark, New Jersey
  - Therapeutics Concepts, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Treon SP, Kotton CN, Park DJ, Moranzoni G, Lemvigh CK, Gathe JC Jr, Varughese TA, Barnett CF, Belenchia JM, Clark NM, Farber CM, Abid MB, Ahmed G, Patterson CJ, Guerrera ML, Soumerai JD, Chea VA, Carulli IP, Southard J, Li S, Wu CJ, Livak KJ, Holmgren E, Kim P, Shi C, Lin H, Ramakrishnan V, Ou Y, Olszewski S, Olsen LR, Keskin DB, Hunter ZR, Tankersley C, Zimmerman T, Dhakal B. A randomized, placebo-controlled trial of the BTK inhibitor zanubrutinib in hospitalized patients with COVID-19 respiratory distress: immune biomarker and clinical findings. Front Immunol. 2025 Jan 21;15:1369619. doi: 10.3389/fimmu.2024.1369619. eCollection 2024. PMID 39906744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 participants were randomized to receive zanubrutinib or placebo; four were randomized to the placebo group, but did not receive placebo treatment due to death (1 participant) and investigator decision (3 participants).
Groups:
- Zanubrutinib + Supportive Care: Zanubrutinib 320 mg orally once daily for 28 days. Supportive care treatment selected and administered as deemed appropriate by the study investigator.
- Placebo + Supportive Care: Placebo orally once daily for 28 days. Supportive care treatment selected and administered as deemed appropriate by the study investigator.
Period: Overall Study
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Started | 30 | 33
Completed | 13 | 17
Not Completed | 17 | 16
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 11 | 8
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.51) | 56.0 (13.30) | 56.0 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 19
  Not Hispanic or Latino | 16 | 26 | 42
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  Black or African American | 3 | 5 | 8
  White | 19 | 25 | 44
  Other | 1 | 1 | 2
  Unknown | 3 | 0 | 3
  Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Failure-free Survival
Description: Number of participants with respiratory failure-free survival, defined as not having died or gone into respiratory failure on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Participants | 27 | 28
Statistical Analysis 1: Comparison: Zanubrutinib + Supportive Care vs Placebo + Supportive Care; Test type: Superiority; p = 0.4099, Unstratified 1-sided Fisher's exact test; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.349 to 7.391]

2. Primary Outcome: Time to Breathing Room Air
Description: Time to return to breathing room air is defined as the time from randomization date to the earliest time where the participant is stable on room air without supplemental oxygen. Total follow-up time in days is the total time of all participants from the randomization date to the first event date or Day 28 if there is no event. The rate was calculated as total number of events in which a participant returned to breathing room air on or before Day 28 divided by the total follow-up time in days.
Time Frame: Up to 7 months
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Number; unit: Events / total follow-up in days
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Events / total follow-up in days | 0.060 | 0.061
Statistical Analysis 1: Comparison: Zanubrutinib + Supportive Care vs Placebo + Supportive Care; Test type: Superiority; p = 0.7619, Log Rank; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.511 to 1.648]

3. Secondary Outcome: Number of Participants Experiencing Respiratory Failure or Death
Description: Number of participants experiencing respiratory failure or death on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Participants | 3 | 5

4. Secondary Outcome: Number of Participants With All-cause Mortality
Description: Number of participants with all-cause mortality on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Participants | 2 | 4

5. Secondary Outcome: Number of Participants Discharged Alive
Description: Number of participants discharged alive on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Participants | 26 | 28

6. Secondary Outcome: Number of Participants Discharged Alive From the ICU
Description: Number of participants discharged alive from the intensive care unit (ICU) on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants; Here, overall number of participants analyzed represents participants who were admitted to the ICU and are evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 14 | 13
Participants | 3 | 2

7. Secondary Outcome: Number of Participants With Improvement in the World Health Organization (WHO) 8-point Ordinal Scale
Description: Number of participants with improvement in WHO 8-point-scale, in which improvement was considered a score that changed from ≥4 at baseline to ≤ 3 at Day 28 as assessed by the investigator. Scoring ranges from 0 = uninfected with no clinical or virologic evidence of disease to 8 = dead.
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Participants | 22 | 25

8. Secondary Outcome: Duration of Mechanical Ventilation
Description: Number of days on mechanical ventilation on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants, excluding participants who died before event completion; Here, overall number of participants analyzed represents participants who progressed from supplemental oxygen to mechanical ventilation and are evaluable for this outcome measure
Measure: Median (Full Range); unit: Days
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 3 | 4
Days | 4.0 [3 to 24] | 13.5 [3 to 26]

9. Secondary Outcome: Duration of Hospitalization
Description: Number of days hospitalized on or before Day 28
Time Frame: Up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants, excluding participants who died before event completion
Measure: Median (Full Range); unit: Days
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 33
Days | 6.5 [3 to 28] | 5.0 [1 to 28]

10. Secondary Outcome: PaO2:FiO2 Ratio
Description: Partial pressure of oxygen (PaO2):fraction of inspired oxygen (FiO2) ratio
Time Frame: Baseline, Day 7, Day 14, Day 21 and Day 28
Population: The Intent-to-Treat Analysis Set included all randomized participants; Here, overall number of participants analyzed represents participants who progressed from supplemental oxygen to mechanical ventilation and are evaluable for this outcome measure and number analyzed represents participants with evaluable data at each time point
Measure: Median (Full Range); unit: mmHg
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 3 | 3
mmHg
  Baseline: number analyzed (Participants) | 0 | 1
  Baseline |  | 53.0 [53.0 to 53.0]
  Day 7: number analyzed (Participants) | 2 | 3
  Day 7 | 82.00 [75.00 to 89.00] | 54.00 [52.80 to 84.30]
  Day 14: number analyzed (Participants) | 1 | 1
  Day 14 | 32.00 [32.00 to 32.00] | 90.60 [90.60 to 90.60]
  Day 21: number analyzed (Participants) | 0 | 1
  Day 21 |  | 52.10 [52.10 to 52.10]
  Day 28: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), treatment-related adverse events (AEs), and TEAEs grade 3 or higher, including laboratory findings
Time Frame: Up to 7 months
Population: The Safety Analysis Set includes all participants who received any dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 30 | 29
Participants
  At least one TEAE | 19 | 20
  Grade 3 or higher | 6 | 6
  Serious adverse event | 4 | 7
  Treatment-related TEAE | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Serious and other (not including serious) adverse events are reported for the Safety Analysis Set, which includes all participants who received any dose of study drug. All-cause mortality is reported for all randomized participants.
Arm/Group | Zanubrutinib + Supportive Care | Placebo + Supportive Care
All-Cause Mortality (participants affected / at risk) | 3/30 | 4/33
Serious Adverse Events (participants affected / at risk) | 4/30 | 7/29
Other Adverse Events (participants affected / at risk) | 19/30 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanubrutinib + Supportive Care (N=30) | Placebo + Supportive Care (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanubrutinib + Supportive Care (N=30) | Placebo + Supportive Care (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 5 (5) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT04382586/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT04382586/SAP_001.pdf